CLINICAL TRIAL: NCT00870298
Title: Randomized Controlled Study of a Computer Stop Order Versus Routine Practice When Trimethoprim/Sulfamethoxazole is Ordered Concurrently With Warfarin
Brief Title: Computer Stop Order Alert to Prevent Concurrent Prescribing of Trimethoprim/Sulfamethoxazole and Warfarin
Acronym: warf-tmp/smx
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: four adverse events encountered
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 803788
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Prescribers' Drug Orders
Keywords: drug orders
MeSH Terms: interventions — Trimethoprim; Sulfamethoxazole; Warfarin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- computerized alert (Experimental): An automatic electronic stop of the tmp/sulfa or warfarin order whenever a resident or nurse practitioner places an order for tmp/sulfa with an already active warfarin order, or when ordering both simultaneously
  Interventions: Drug: Trimethoprim/Sulfamethoxazole and Warfarin
- 2 Current practice (Other): Current practice of the pharmacist recommending cessation of concurrent warfarin and tmp/sulfa orders
  Interventions: Drug: Trimethoprim/Sulfamethoxazole and Warfarin

INTERVENTIONS:
Drug: Trimethoprim/Sulfamethoxazole and Warfarin

SUMMARY:
To determine if a computerized stop order will reduce the number of concurrent trimethoprim/sulfamethoxazole and warfarin orders accepted through the inpatient electronic ordering system while a patient is hospitalized.

ELIGIBILITY:
Inclusion Criteria:

All resident physicians and nurse practitioners involved in inpatient care.

Exclusion Criteria:

None-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1971 (Actual)
Dates: Start 2006-08; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Reduce concomitant orders for warfarin and tmp/smx | 7 months

SECONDARY OUTCOMES:
Determine if computerized stop order will increase risk for inadvertent cessation of warfarin | 7 months
Determine if computerized stop order will increase risk of delay of treatment with tmp/sulfa when determined to be necessary for treatment | 7 months

REFERENCES:
- [Derived] Strom BL, Schinnar R, Aberra F, Bilker W, Hennessy S, Leonard CE, Pifer E. Unintended effects of a computerized physician order entry nearly hard-stop alert to prevent a drug interaction: a randomized controlled trial. Arch Intern Med. 2010 Sep 27;170(17):1578-83. doi: 10.1001/archinternmed.2010.324. PMID 20876410